CLINICAL TRIAL: NCT03416478
Title: The Implication of Plasma Circulating Tumor DNA (ctDNA) in the Recurrence Surveillance of Stage II and III Colorectal Cancer: a Prospective Study
Brief Title: The Implication of ctDNA in the Recurrence Surveillance of Stage II and III Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaojian Wu, Vice President, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: FFJC2017-01
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer; ctDNA; Surveillance
Keywords: Colorectal Cancer; ctDNA; Surveillance
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ctDNA test group
  Interventions: Diagnostic Test: ctDNA test

INTERVENTIONS:
Diagnostic Test: ctDNA test — ctDNA test to find some possible mutation.

SUMMARY:
This study is to evaluate circulating tumor DNA (ctDNA) as a predictive and surveillant method for tumor recurrence in stage II and III colorectal cancer (CRC).

DETAILED DESCRIPTION:
This study will evaluate circulating tumor DNA (ctDNA) as a prognostic marker and as a monitor of a short-term disease recurrence in surgical resective stage II and stage III colorectal cancer (CRC). The investigators will recruit newly diagnosed CRC patients, systematically collect their blood samples at the following time point: before surgery, one week after surgery, every three months for the first year and every six months for the second year, which are coincidence with the recommended clinical follow-up. Patients' outcome and survival will be tracked. These study will permit assessment of ctDNA as a predictive and surveillant method for a short-term (two years) tumor recurrence in comparison with other parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age on the day of signing informed consent.
* Patients must have histologically confirmed stage II or IIIcolorectal cancer.
* Patients must receive radical resection.
* Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

* Patient has severe anemia.
* Patients received neoadjuvant treatment.
* Patients received blood transfusion two weeks before or during the surgical resection.
* Patient has any other conditions, which, in the opinion of the Investigator, would interfere with the evaluation of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II or stage III colorectal cancer must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | Two years

SECONDARY OUTCOMES:
Overall survival | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojian Wu, MD, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yet-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yet-sen University, Guangzhou, China